CLINICAL TRIAL: NCT00132314
Title: CSP #555 - Long-Acting Injectable Risperidone in the Treatment of Schizophrenia
Brief Title: Long-Acting Injectable Risperidone in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 555
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-10

CONDITIONS: Schizoaffective Disorder; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): long-acting injectable risperidone
  Interventions: Drug: IM risperidone
- Arm 2 (Active Comparator): oral antipsychotic medication
  Interventions: Drug: oral antipsychotic medication

INTERVENTIONS:
Drug: IM risperidone — long-acting injectable risperidone
  Arms: Arm 1
Drug: oral antipsychotic medication — doctor's choice (excluding other long-acting injectable medications but not specifying any particular oral agents or dosages)
  Arms: Arm 2

SUMMARY:
In the proposed study 450 veterans with a primary diagnosis of schizophrenia who had at least one psychiatric hospitalization for schizophrenia in the previous 2 years would be randomly assigned at 16 VA medical centers to long-acting injectable risperidone or doctor's choice of oral antipsychotic medication (i.e., excluding other long-acting injectable medications, but not specifying any particular oral agents or dosages). Recruitment would take 27 months to complete, and the study would continue for a third year to allow 9 months of follow-up for the last patient recruited. All patients would be treated from the time of entry up to the end of the three-year study period. Follow-up assessments would continue quarterly. Treatments would not be blinded since giving placebo injections to the comparison group would interfere with the goal of comparing the acceptability of two different methods of medication administration. However, end points will be blindly rated.

DETAILED DESCRIPTION:
The purpose of the study is to assess the effectiveness of long-acting injectable risperidone on psychiatric inpatient hospitalization, schizophrenia symptoms, quality of life, medication adherence, side effects, and health care costs.

Objectives:

Primary: To evaluate the impact of long-acting intramuscular (IM) risperidone on risk of inpatient psychiatric hospitalization in comparison to standard oral antipsychotic treatment in a randomized controlled trial to be conducted with 450 veterans diagnosed with schizophrenia or schizoaffective disorder at 16 VA medical centers over three years.

Secondary: To evaluate adherence, health benefits, and costs of long-acting IM risperidone as compared to standard oral antipsychotic treatment as measured by: a) symptom reduction over 12 months, b) time to all-cause medication discontinuation, c) quality of life, d) VA and non-VA health service use and related costs, e) medication side effects, f) violent behavior, g) use of concomitant medication, and h) the incremental cost-effectiveness ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosed with schizophrenia or schizoaffective disorder by the Structured Clinical Interview for Diagnosis (SCID) (Spitzer and First et al., 1996).
3. Patients should

   1. have been hospitalized in the two years before study entry on a psychiatric inpatient unit, or
   2. document explicit current evidence of increased use of outpatient services such as additional visits, day treatment or non-hospital residential treatment, increased dosage of medications or addition of concomitant psychotropic medications.

   The b criterion will promptly be adjudicated by the study chairmen on a case-by case basis to insure credibility.
4. .Adequate transportation is available and the participant lives within a travel time of less than 1.5 hours, allowing attendance at all scheduled visits.
5. Use of an acceptable method of birth control by female patients who have a possibility of becoming pregnant (safety concerns).
6. Able to demonstrate decisional capacity in order to give informed consent as assessed by the MacArthur Competence Assessment Tool (MacCAT) (Appelbaum and Grisso, 1996). Guardian consent is acceptable where applicable.
7. Dually diagnosed patients with both schizophrenia and addictive disorders would be included in this study but should not be in need of acute detoxification for physiologic substance dependence (excluding nicotine) in the past 30 days.

Exclusion Criteria:

1. Physiologic substance dependence requiring detoxification (excluding nicotine) in the past 30 days (substance abuse is not an exclusion).
2. Intolerance of risperidone.
3. Intolerance of intramuscular injection.
4. Current treatment with depot antipsychotic medication.
5. Current treatment with oral clozapine or presence of refractory schizophrenia that, in the treating psychiatrist's opinion, requires clozapine.
6. Hepatic or renal problems AST or ALT (>2 times upper limit of normal);
7. Elevated bilirubin (>1.2), BUN (>24), creatinine (>1.7).
8. Unstable, serious medical condition or one requiring acute medical treatment, or anticipation of hospitalization for extended care.
9. Dementia, epilepsy, insulin-dependent diabetes, anticoagulation with coumadin.
10. Unstable living arrangements or not planning to remain in the area for the next year.
11. Legal entanglements or pending legal charges with potential of incarceration.
12. Assault or suicide gesture currently needing acute intervention.
13. Concurrent participation in another clinical trial with an investigational drug during the last 30 days.
14. Pregnant or lactating women or women planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Rosenheck, AB MD, Study Chair — VA Connecticut Health Care System (West Haven)
Locations (19):
- United States (19):
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Miami, Miami, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, Omaha, Omaha, Nebraska
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Central Texas Veterans Health Care System - Waco, Waco, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Rosenheck RA, Krystal JH, Lew R, Barnett PG, Thwin SS, Fiore L, Valley D, Huang GD, Neal C, Vertrees JE, Liang MH; CSP 555 Research Group. Challenges in the design and conduct of controlled clinical effectiveness trials in schizophrenia. Clin Trials. 2011 Apr;8(2):196-204. doi: 10.1177/1740774510392931. Epub 2011 Jan 26. PMID 21270143
- [Result] Rosenheck RA, Krystal JH, Lew R, Barnett PG, Fiore L, Valley D, Thwin SS, Vertrees JE, Liang MH; CSP555 Research Group. Long-acting risperidone and oral antipsychotics in unstable schizophrenia. N Engl J Med. 2011 Mar 3;364(9):842-51. doi: 10.1056/NEJMoa1005987. PMID 21366475
- [Result] Barnett PG, Scott JY, Rosenheck RA; CSP 555 Study Group. How do clinical trial participants compare to other patients with schizophrenia? Schizophr Res. 2011 Aug;130(1-3):34-9. doi: 10.1016/j.schres.2011.03.033. Epub 2011 Apr 22. PMID 21514794
- [Result] Barnett PG, Scott JY, Krystal JH, Rosenheck RA; CSP 555 Research Group. Cost and cost-effectiveness in a randomized trial of long-acting risperidone for schizophrenia. J Clin Psychiatry. 2012 May;73(5):696-702. doi: 10.4088/JCP.11m07070. PMID 22697193
- [Result] Thwin SS, Hermes E, Lew R, Barnett P, Liang M, Valley D, Rosenheck R. Assessment of the minimum clinically important difference in quality of life in schizophrenia measured by the Quality of Well-Being Scale and disease-specific measures. Psychiatry Res. 2013 Oct 30;209(3):291-6. doi: 10.1016/j.psychres.2013.01.016. Epub 2013 Mar 7. PMID 23473656
- [Derived] Hoblyn JC, Rosenheck RA, Leatherman S, Weil L, Lew R; CSP 555 Investigator Group. Veteran subjects willingness to participate in schizophrenia clinical trials. Psychiatr Q. 2013 Jun;84(2):209-18. doi: 10.1007/s11126-012-9240-4. PMID 23143523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2006 - December 2008; 19 VA medical centers
Groups:
- Injectable Risperidone: long-acting injectable risperidone
- Oral Antipsychotic: oral antipsychotic medication
Period: Overall Study
Arm/Group | Injectable Risperidone | Oral Antipsychotic
Started | 190 | 192
Received Treatment | 188 | 185
Completed Baseline Visit, Provided SSN | 187 (This is the ITT cohort) | 182 (This is the ITT cohort.)
Completed | 117 | 120
Not Completed | 73 | 72
Not completed — Lost to Follow-up | 70 | 62
Not completed — Lacked SSN | 1 | 3
Not completed — Refused intervention at baseline | 2 | 7

BASELINE CHARACTERISTICS:
Population: We used the intention to treat (ITT) population as defined in Milestone 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectable Risperidone | Oral Antipsychotic | Total
Number analyzed (Participants) | 187 | 182 | 369
Age Continuous [Mean (Standard Deviation); unit: years] | 50.6 (9.7) | 51.3 (8.8) | 50.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 172 | 165 | 337

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization-free Survival - Time to Event
Description: A hospitalization-free survival was defined as the time from the date of randomization to the time of a psychiatric hospitalization (in both VA and non-VA hospitals) or, in the case of patients who were hospitalized at randomization, the time from the date of discharge from the initial stay to subsequent hospitalization. Patients without an event were censored at 24 months after the date of randomization.
Time Frame: From randomization until date of first re-hospitalization, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Injectable Risperidone | Oral Antipsychotic
Number analyzed (Participants) | 187 | 182
years | NA [1.84 to NA] — The median time to event based on Kaplan-Meier estimates was not reached, and upper 95% confidence interval could not be estimated | 1.97 [1.19 to NA] — Upper 95% confidence interval could not be estimated
Statistical Analysis 1: Comparison: Injectable Risperidone vs Oral Antipsychotic; Time-to-event analysis; The primary outcome hypothesis is tested using a two-sided log-rank test to compare the hazard rate for the IM treatment group to that for the oral treatment group; Test type: Superiority or Other; p = 0.39, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.63 to 1.20]

2. Primary Outcome: Hazard Ratio for Hospitalization
Description: Hazard ratio of LAI versus Oral for psychiatric hospitalization (in both VA and non-VA hospitals), after randomization up to 24 months, obtained from a Cox proportional hazards model.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Injectable Risperidone | Oral Antipsychotic
Number analyzed (Participants) | 187 | 182
participants
  Patients with psychiatric hospitalization | 72 | 81
  Patients without psychiatric hospitalization | 115 | 101
Statistical Analysis 1: Comparison: Injectable Risperidone vs Oral Antipsychotic; Test type: Superiority or Other; Regression, Cox — 95% Confidence Interval: 0.63 to 1.20; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.63 to 1.20]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to 30 days after the end of follow-up. Subjects were followed for up to 36 months, depending on when the participant was enrolled in the study.
Description: Participants were monitored for adverse events (AEs) and serious adverse events (SAEs) at monthly study visits. AEs and SAEs were both actively and passively monitored.
Arm/Group | Injectable Risperidone | Oral Antipsychotic
Serious Adverse Events (participants affected / at risk) | 96/187 | 91/182
Other Adverse Events (participants affected / at risk) | 132/187 | 123/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectable Risperidone (N=187) | Oral Antipsychotic (N=182)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (4)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (5) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Anticonvulsant drug level increased (Investigations) | 1 (1) | 0 (0)
Antipsychotic drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Sedation (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Tardive dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 7 (7) | 8 (10)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 47 (87) | 56 (104)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 37 (51) | 38 (63)
Suicide attempt (Psychiatric disorders) | 4 (4) | 9 (9)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug abuser (Social circumstances) | 1 (1) | 0 (0)
Substance abuse (Social circumstances) | 1 (1) | 1 (1)
Drug detoxification (Surgical and medical procedures) | 2 (2) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Pleural decortication (Surgical and medical procedures) | 1 (1) | 0 (0)
Radical prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectable Risperidone (N=187) | Oral Antipsychotic (N=182)
Vertigo (Ear and labyrinth disorders) | 21 (26) | 22 (28)
Vision blurred (Eye disorders) | 10 (10) | 12 (14)
Constipation (Gastrointestinal disorders) | 22 (33) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 13 (15)
Dry mouth (Gastrointestinal disorders) | 21 (34) | 22 (29)
Salivary hypersecretion (Gastrointestinal disorders) | 13 (16) | 7 (10)
Vomiting (Gastrointestinal disorders) | 26 (34) | 24 (34)
Chest pain (General disorders) | 10 (15) | 9 (10)
Fatigue (General disorders) | 24 (29) | 23 (32)
Nasopharyngitis (Infections and infestations) | 13 (19) | 11 (13)
Weight increased (Investigations) | 14 (15) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 13 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (13) | 5 (5)
Akathisia (Nervous system disorders) | 22 (28) | 12 (13)
Extrapyramidal disorder (Nervous system disorders) | 14 (21) | 9 (9)
Headache (Nervous system disorders) | 32 (44) | 25 (35)
Sedation (Nervous system disorders) | 13 (14) | 16 (17)
Insomnia (Psychiatric disorders) | 35 (52) | 44 (60)
Dysuria (Renal and urinary disorders) | 10 (13) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 18 (26) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No